CLINICAL TRIAL: NCT07056829
Title: The Effect of Mandibular Advancement With Clear Aligners on Maxillary and Mandibular Volumes: A Randomized Controlled Trial Using CBCT
Brief Title: The Effect of Mandibular Advancement With Clear Aligners on Maxillary and Mandibular Volumes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batman University (Other)
Responsible Party: Principal Investigator, Nursezen Kavasoglu, Assistant Professor Dr., Batman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NK02
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Mandibular Retrognathia
Keywords: clear aligners; mandibular retrognathia; mandibular advancement
MeSH Terms: conditions — Micrognathism | interventions — Activator Appliances

STUDY DESIGN:
Intervention Model Description: This study follows a parallel assignment model. Participants are randomly assigned to one of three groups: the Mandibular Advancement Appliance (MAA) group, the Activator group, or the control group. Each group receives a different intervention or, in the case of the control group, no treatment, and all groups are observed over the same period without crossover between interventions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MAA Group (Experimental): Patients receive orthodontic treatment using clear aligners (Invisalign) with integrated mandibular advancement features (MAA). Advancement is performed in 2 mm increments every 8 weeks over ~8 months.
  Interventions: Device: Mandibular Advancement Appliance (Invisalign MA)
- Activator Group (Active Comparator): Patients receive traditional removable functional appliance therapy (Activator) for ~7 months.
  Interventions: Device: Activator Appliance
- Control Group (No Intervention): Patients receive no orthodontic treatment but are monitored for the same duration as the treatment groups.

INTERVENTIONS:
Device: Mandibular Advancement Appliance (Invisalign MA) — Clear aligner system with integrated buccal precision wings to posture the mandible forward.
  Advancement protocol: 2 mm increments every 8 weeks. Total active treatment duration: ~8.15 months, followed by retention phase. Patients instructed to wear aligners ≥20 h/day, removing only for eating and oral hygiene.
  Arms: MAA Group
Device: Activator Appliance — Traditional removable functional appliance fabricated on a standardized bite registration.
  Patients instructed to wear appliance 24 h/day except during meals and sports. Total active treatment duration: ~7.15 months, followed by retention phase.
  Arms: Activator Group

SUMMARY:
The aim of this study is to compare the effectiveness of two different orthodontic treatment methods used in patients with skeletal Class II malocclusion, a condition in which the lower jaw is positioned backward. Approximately 80% of Class II malocclusions are due to mandibular retrusion. Therefore, functional appliances that stimulate mandibular growth in growing individuals have been widely used in orthodontics for many years.

In recent years, clear aligner systems have become increasingly popular in orthodontic practice. A mandibular advancement feature was recently integrated into these aligners, allowing for simultaneous tooth alignment and forward positioning of the lower jaw. In this study, the newly developed Mandibular Advancement Appliance (MAA), based on clear aligners, will be compared to the traditional functional appliance known as the Activator.

Who Can Participate in the Study? Children with retrusive lower jaws who are in the growth and development period Individuals with no prior orthodontic treatment Patients with specific levels of dental protrusion (overjet) Those with good general health and no contraindications for CBCT imaging What Will the Treatment Process Involve?

Participants will be randomly assigned to one of three groups:

MAA group (clear aligners with mandibular advancement) Activator group (traditional removable appliance) Control group (no treatment, only observation) The active treatment period will last approximately 7-8 months, followed by a retention phase. All patients will be monitored regularly, and strict adherence to appliance use will be expected.

How Will the Outcomes Be Assessed? Before and after the treatment period, participants will undergo cone-beam computed tomography (CBCT) scans to obtain detailed three-dimensional images of the jaws. These images will be analyzed to evaluate volumetric changes. All measurements will be performed by a trained orthodontic specialist using dedicated software.

Potential Benefits for Participants:

Participants will receive close clinical monitoring throughout the study period. The use of advanced imaging technologies may support the development of more effective and individualized treatment plans.

Safety and Confidentiality:

This study has received ethical approval and will be conducted in accordance with relevant data protection and research ethics standards. All personal data will be kept confidential. Written informed consent will be obtained from all participants and/or their legal guardians.

ELIGIBILITY:
Inclusion Criteria:

* Cervical vertebral maturation (CVM) stage 2 or 3
* Bilateral full or half cusp Class II molar relationship
* Skeletal Class II relationship associated with mandibular retrognathia (ANB angle > 4° and SNB angle < 78°)
* Horizontal or average growth pattern (SN-GoGn ≤ 38°)
* Overjet distance between +4 mm and +8 mm; (6) Good patient compliance throughout the treatment.

Exclusion Criteria:

* CVM stage 5 or 6;(2) Previous orthodontic treatment;
* Presence of maxillary prognathism
* High-angle growth pattern (SN-GoGn > 38°)
* Transverse orthodontic anomalies or facial asymmetry
* Palpation-induced tenderness or pain in the masticatory muscles
* Presence of clicking, crepitus, pain, or tenderness in the temporomandibular joint (TMJ)
* Congenital or acquired craniofacial deformities
* Poor patient compliance or oral hygiene
* Any condition that could interfere with CBCT imaging.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Change in mandibular volume (mm³) | Baseline and post-treatment (~8 months)
  Mandibular volume change will be measured using CBCT scans analyzed via Mimics software. The MAA and Activator groups will be compared to evaluate treatment effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Batman University Faculty of Dentistry, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No